CLINICAL TRIAL: NCT07180875
Title: Simulated Hypoxia Training to Enhance Exercise Tolerance in Stage 3 Chronic Kidney Disease: A Randomized Controlled Trial
Brief Title: "Hypoxic vs. Aerobic Training in Chronic Kidney Disease
Acronym: IHT-CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, ola mohamed elgohary, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OlaElgohary-IHT-CKD-01
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease (CKD), Stages 3-4 Exercise Tolerance / Functional Capacity Vascular Health / Arterial Stiffness Fatigue in CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking Description: Outcome assessors and data analysts will be blinded to group allocation; participants and trainers cannot be blinded due to the nature of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypoventilation Training group (Experimental): * Mode: Stationary cycling (ergometer).
  * Intensity: Moderate (40-60% VO₂max or Borg RPE 11-13).
  * Duration: 30 minutes per session.
  * Frequency: 3 sessions per week, for 12 weeks.
  * Technique:
    * Patients instructed to hold their breath (hypoventilation) for 5-10 seconds every 2-3 minutes during cycling.
    * Breathing then resumes normally until recovery.
    * Cycle repeated throughout the session
  Interventions: Behavioral: hypoventilation group
- Breathing Restriction Mask Training (Experimental): * Mode: Stationary cycling (ergometer).
  * Intensity: Moderate (same as Group A: 40-60% VO₂max).
  * Duration: 30 minutes per session.
  * Frequency: 3 sessions per week, for 12 weeks.
  * Equipment: Commercially available breathing restriction mask (e.g., altitude simulation mask).
  * Technique:
    * Mask settings adjusted to provide increasing resistance over time, simulating hypoxic breathing (FiO₂ ~14-16%).
    * Patients cycle continuously with mask worn throughout the session.
  * Monitoring:
    * SpO₂, HR, BP monitored continuously.
    * Mask removed immediately if SpO₂ < 88% or severe dyspnea occurs.
  Interventions: Behavioral: hypoventilation group
- Control Group (Conventional Aerobic Training) (Active Comparator): * Mode: Stationary cycling (ergometer).
  * Intensity: Moderate (40-60% VO₂max or Borg RPE 11-13).
  * Duration: 30 minutes per session.
  * Frequency: 3 sessions per week, for 12 weeks.
  * Technique:
    * Continuous cycling at steady pace.
    * No hypoventilation or mask used.
  * Monitoring:
    o HR, BP, and SpO₂ checked pre- and post-session.
  * Progression:
    * Workload (watts) increased every 2-3 weeks to maintain moderate intensity
  Interventions: Behavioral: hypoventilation group

INTERVENTIONS:
Behavioral: hypoventilation group — Traditional Aerobic Training Participants will perform supervised aerobic exercise (e.g., cycling or treadmill walking) under controlled intermittent hypoxic conditions.
  Hypoxia protocol: alternating cycles of low-oxygen exposure (FiO₂ 12-16%) for 3-5 minutes followed by normoxic recovery for 2-3 minutes, repeated 6-8 times per session.
  Frequency: 3 sessions per week for 12 weeks.
  Exercise intensity: Moderate (50-70% of heart rate reserve), adjusted individually based on baseline exercise testing
  Other Names: Breathing Restriction Mask Training

SUMMARY:
Chronic kidney disease (CKD) leads to poor exercise tolerance, vascular dysfunction, and reduced quality of life. This randomized controlled trial will compare intermittent hypoxic training (IHT) with traditional aerobic training in patients with CKD stages 3-4.

A total of 60 participants aged 40-65 years will be recruited and randomized into three groups. Interventions will last 12 weeks, with three 30-minute supervised sessions per week. Outcome measures include exercise tolerance (6-Minute Walk Test), cardiovascular parameters (blood pressure, heart rate recovery), kidney function (serum creatinine, eGFR), fatigue (Fatigue Severity Scale), and quality of life (KDQOL-36)

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) stage 3 is characterized by reduced exercise capacity, muscle weakness, and increased cardiovascular risk, which negatively impact quality of life. Exercise interventions have shown benefits in improving functional outcomes, but traditional aerobic training may be limited due to comorbidities and reduced physiological reserve. Intermittent hypoxic training (IHT) improves oxygen utilization, cardiovascular adaptation, and mitochondrial function. Specialized hypoxicator devices are costly and not widely available, so practical alternatives such as hypoventilation training and breathing restriction masks may provide comparable benefits.

Study Objective:

To evaluate the effects of hypoventilation training and breathing restriction mask training on exercise tolerance, cardiovascular function, kidney function, fatigue, and quality of life in CKD stage 3 patients.

Study Design:

Randomized controlled trial including 60 patients with CKD stage 3, aged 40-65 years, recruited from outpatient clinics at Aboker Hospital and Pharos University. Participants will be screened for eligibility through medical history, vital signs, and laboratory tests (serum creatinine, eGFR, hemoglobin, electrolytes).

Interventions:

Group A - Hypoventilation Training:

Moderate-intensity aerobic exercise on a cycle ergometer (40-60% HR reserve)

Intermittent breath-holding: 5-10 seconds every 1-2 minutes

Continuous monitoring of SpO₂, heart rate, and blood pressure

Group B - Breathing Restriction Mask Training:

Same aerobic protocol as Group A

Participants wear an adjustable resistance mask to simulate hypoxia

Mask set to induce mild hypoxemia (SpO₂ ≥85%)

Continuous monitoring of SpO₂, heart rate, and blood pressure

Group C - Control Group:

Same aerobic exercise protocol under normal breathing conditions

Moderate intensity (40-60% HR reserve)

Periodic monitoring of vital signs for safety

Intervention Duration:

12 weeks, 3 supervised sessions per week, 30 minutes per session

Outcome Measures:

Primary Outcome:

Exercise tolerance assessed via 6-Minute Walk Test (6MWT) at baseline and post-intervention

Secondary Outcomes:

Fatigue: Fatigue Severity Scale (FSS), self-reported, 9 items, 7-point Likert scale

Quality of Life: KDQOL-36, disease-specific questionnaire covering physical/mental health, symptoms, effects, and burden of CKD

Cardiovascular Assessment: Blood pressure (SBP, DBP) and Heart Rate Recovery (HRR = HR_peak - HR_1min)

Kidney Function: Serum creatinine and eGFR (CKD-EPI/MDRD

ELIGIBILITY:
Inclusion Criteria:Adults (40-65 years) diagnosed with CKD stages 3a,b

* Medically stable and cleared for exercise

Exclusion Criteria:

* Uncontrolled hypertension
* Severe cardiac arrhythmias
* Recent hospitalization (<3 months)

cardiovascular disese unstable

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both men and women are eligible; no gender restriction
Enrollment: 60 (Estimated)
Dates: Start 2025-12-09 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test (6MWT) distance | 12 weeks
  Straightforward standardized 6-minute corridor walk performed according to ATS guidelines. Participants walk back and forth along a marked 30-meter course for 6 minutes; standardized instructions and encouragement are given. Total distance walked (meters) recorded. Assessors are blinded to group allocation.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 12 wwks
  A validated 9-item self-report questionnaire assessing the impact and severity of fatigue on daily functioning. Each item is rated on a 7-point Likert scale; higher scores indicate greater fatigue.
Kidney Disease Quality of Life Questionnaire (KDQOL-36) | 12 weeks
  A disease-specific quality of life tool combining general health status (SF-12) and kidney disease-targeted domains (symptoms/problems, effects, and burden of kidney disease). Scores are standardized (0-100), with higher scores indicating better quality of life

IPD SHARING:
Plan to Share IPD: Undecided
This study will compare the effects of intermittent hypoxic training (IHT) versus traditional aerobic training (TAT) on exercise tolerance and vascular health in patients with chronic kidney disease (CKD) stages 2-4. Participants will be randomized into two intervention groups and undergo supervised exercise sessions over a 12-week period. Primary outcomes include peak oxygen uptake (V̇O₂peak) and endothelial function (flow-mediated dilation), while secondary outcomes include arterial stiffness, 6-minute walk distance, and quality of life measures. Safety and adherence will be closely monitored throughout the study. Data will be analyzed to determine the comparative efficacy of IHT and TAT in improving functional and vascular health in this population